CLINICAL TRIAL: NCT04971044
Title: COACH: Competency Based Approaches for Community Health 2
Brief Title: Competency Based Approaches for Community Health 2
Acronym: COACH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of North Carolina, Chapel Hill (Other); Vanderbilt University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Bill Heerman, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R01HD100458 (NIH); 3R01HD100458-03S1 (NIH)
Record Dates: First submitted 2020-10-26; First posted 2021-07-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Obesity
Keywords: Childhood Obesity; Behavioral Intervention; Parent-Child Pairs; Low-Income, Minority Populations; Hispanic/Latino Populations
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COACH Intervention (Experimental): COACH is a multi-level intervention, consisting of 1) developmentally appropriate health curriculum for 4-6 year old children; 2) family-based content that both targets parent weight loss and leverages a shared parent-child experience to improve family health behaviors; 3) community-level intervention to improve access and quality of family-based programming at local Parks and Rec centers.
  Interventions: Behavioral: COACH
- Educational Control (Active Comparator): The control arm will consist of a school readiness intervention developed by education and literacy experts on our team and implemented at local libraries. It will include 1) child lessons from Puente de Cuentos, a systematic, language-based curriculum focused on dual language storytelling (narrative language), and 2) parent sessions designed to improve parents' knowledge and skills related to improving children's language production and storytelling skills, to ultimately support school readiness.
  Interventions: Behavioral: School Readiness Intervention

INTERVENTIONS:
Behavioral: COACH — Multi-Level Behavioral Intervention
  Arms: COACH Intervention
Behavioral: School Readiness Intervention — Multi-Level Language and School Readiness Intervention (Control Group)
  Arms: Educational Control

SUMMARY:
One-size-fits-all approaches have failed to demonstrate sustained effects on childhood obesity, especially among low-income minority families, who experience constantly changing barriers to engaging in health behavior. Addressing obesity in these populations requires intervening in early childhood and situating interventions in the context of families and communities. Developing personalized childhood obesity prevention interventions with sustained effectiveness that support families in health behaviors despite dynamic barriers could address chronic disease risk and health disparities in low-income and minority communities.

DETAILED DESCRIPTION:
Despite the recognition of health disparities in obesity, behavioral interventions among low-income and minority populations have consistently met with limited success. This is partially explained by social determinants of health. Constantly changing barriers at the household and community levels impede consistent engagement in healthy behaviors. The current proposal tests a novel, culturally-tailored and multi-level intervention designed to teach families to overcome dynamic barriers as the logical next step to address obesity among low-income Latino families. It is based on the premise that by implementing a personalized multi-level intervention that simultaneously addresses healthy weight for parents and children, we will improve body mass index (BMI) among Latino parent-child pairs.

COACH (COmpetency-Based Approaches to Community Health) implements a personally tailored approach, equipping families to engage in health behaviors despite dynamic barriers. COACH is a multi-level intervention targeting 1) the individual child through developmentally appropriate health behavior curriculum, 2) the family by addressing parent weight loss directly and engaging parents as agents of change for their children, and 3) the community by building capacity of Parks and Rec centers to offer parent-child programming. Using novel multi-component assessments throughout the study, the intervention identifies individual, family, and community barriers to healthy behaviors and delivers structured yet personalized intervention content in 7 domains: fruits/vegetables, snacks, sugary drinks, physical activity, sleep, media use, and parenting.

Building on a successful pilot, this proposal will implement a randomized controlled trial to test the effectiveness of COACH compared to an attention-matched school-readiness control group. We will enroll 300 parent-child pairs from Latino communities in Nashville, TN.

The goals of COACH are to 1) implement a novel personalized behavioral intervention, 2) test a two-generation solution to obesity, 3) address health disparities by reducing obesity among Latino families, and 4) develop a scalable and widely accessible approach to behavioral obesity interventions by delivering them in Parks and Rec centers.

ELIGIBILITY:
Inclusion Criteria:

* child with an age ≥4 years and <7 years;
* index parent/legal guardian with an age ≥18 years;
* English- or Spanish-speaking;
* self-identify as Hispanic/Latino;
* live in a home where Spanish is spoken;
* include an index parent/legal guardian with a body mass index of ≥25kg/m2 and <55 kg/m2;
* include a child with a body mass index ≥5th percentile percentile for age and gender on standardized CDC growth curves;
* for participants intending to attend intervention sessions in person: reside within or frequent (i.e. work in or regularly visit) one of the following zip codes: South Nashville/Regions 1 and 2 (37013, 37204, 37210, 37211, 37217, 37220, 37076, 37086, 37167): surrounding the Coleman Recreation Center and Southeast Recreation Center; and Northeast Nashville/Madison/Region 3 (37115, 37138, 37072, 37207, 37216); for participants intending to attend intervention sessions via videoconference: participants may reside in any zip code;
* have parental commitment to participate in a two-year research study;
* have consistent mobile phone access;
* are without medical conditions necessitating limited physical activity as evaluated by a pre-screen;
* complete baseline data collection, including parent and child height and weight and at least 90% of baseline survey items;
* are considered underserved, measured by parent-self reporting that they or someone in their household are eligible for or participate in one of these programs or services: TennCare, CoverKids, WIC, Food Stamps (SNAP), Free and Reduced Price School Lunch and Breakfast, and/or Families First (TANF)

Child exclusion criteria:

* Children outside the specified age range
* Children who are <5th percentile on standardized CDC growth curves
* Children who do not speak English or Spanish
* Children who are diagnosed with medical illnesses where regular exercise might be contraindicated
* Children who display dissenting behaviors during baseline assent or anthropometric data collection
* Children who do not otherwise meet the eligibility criteria listed in section above as determined by pre-screen
* Children who are diagnosed with autism

Caregiver exclusion criteria include:

* Parents/legal guardians who are <18 years old;
* Parents/legal guardians with serious mental or neurologic illness that impairs ability to consent/participate;
* Parents/legal guardians with poor visual acuity (corrected vision worse than 20/50 with Rosenbaum Screener).
* Parents/legal guardians with BMI <25kg/m2 or BMI ≥55kg/m2
* Parents/legal guardians who are diagnosed with medical illnesses where regular exercise might be contraindicated
* Lack of parental commitment to participate consistently for a two-year period
* Lack of telephone contact
* Parents/legal guardians who do not otherwise meet the eligibility criteria listed in section above as determined by pre-screen

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Child Body Mass Index | 24-month follow-up
  Measured prospectively and calculated from child weight/height measures

SECONDARY OUTCOMES:
Parent Body Mass Index | 24-month follow-up
  Measured prospectively and calculated from parent weight/height measures
Child Obesity | 24-month follow-up
  Percent of children with BMI ≥95th percentile on standardized CDC growth curves
Child Overweight | 24-month follow-up
  Percent of children with BMI percentile ≥85th but less than <95th percentile on standardized CDC growth curves
Child Body Mass Index Percentage of the 95th Percentile | 24-month follow-up
  Child BMI percentage of the 95th percentile on standardized CDC growth curves
Child Body Mass Index z-Scores | 24-month follow-up
  Child BMI z-scores on standardized CDC growth reference charts

OTHER OUTCOMES:
Child Diet | 24-month follow-up
  Parent reported diet quality based on survey measures
Parent Diet | 24-month follow-up
  Self-report diet quality based on survey measures
Parent Physical Activity | 24-month follow-up
  Parent reported physical activity for themselves based on survey measures
Child Media Use | 24-month follow-up
  Parent reported media use by child based on survey measures
Child Sleep | 24-month follow-up
  Parent reported sleep times based on survey measures

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
We will plan to upload a de-identified dataset to the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH) database (this upload also includes study protocols).
Supporting Information: Study Protocol, SAP
Time Frame: In accordance with NIH policy, we will make these data available no later than 3 years after the end of the trial (final patient follow-up) or 2 years after the main paper of the trial has been published, whichever comes first.
Access Criteria: Determined by NIH DASH website
URL: https://dash.nichd.nih.gov/